CLINICAL TRIAL: NCT00997529
Title: Nonmyeloablative Allogeneic Stem Cell Transplantation for the Treatment of Solid
Brief Title: Mini Allo Stem Cell Transplantation for the Treatment of Solid Tumors
Acronym: MiniSolid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, David McDermott, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-00-0154-FB/2001-P-000092/8
Record Dates: First submitted 2008-05-05; First posted 2009-10-19 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Solid Tumor
Keywords: Stem cell transplant; Non-myeloablative; Metastatic Solid Tumor; Donor Leukocyte Infusion
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: nonmyeloablative stem cell transplant

INTERVENTIONS:
Drug: nonmyeloablative stem cell transplant — Conditioning includes cytoxan 60mg/kg/d on Days 6 & 5, total dose 120mg/kg, Fludarabine 25mg/m2/d on days -5 to -1, total dose 125mg/m2. Patients with decreased cardiac or liver function pre-transplant will have their dose of cytoxan reduced by 25% - 45 mg/kg/d for 2 days or total dose of 90mg/kg. Patients will receive G-CSF (5ug/kg) to foster engraftment. PBSC progenitors will be mobilized from donor with G-CSF 5ug/kg 2x daily starting 4 days prior to stem cell collection until a target of 5-10 x106 CD34+ cells/kg is reached. Peripheral blood progenitors will be isolated from leukaphereses obtained on Days 5 & 6 with additional collections dependent on cell yields. Peripheral blood from donors will be given to patients 1 day after cytoreduction & immunosuppression. Immunosuppression will be tapered Day +60 if no signs of GVHD. Patients with residual non-regressing disease or mixed chimerism after day 100, who are off immunosuppression & do not have signs of GVHD, will receive a DLI

SUMMARY:
A major focus of recent research has been the development of effective ways of sensitizing the patient's immune system to recognize the cancer as foreign. Allogeneic stem cell transplantation represents a novel way of potentially achieving this goal. There is recent evidence that non-myeloablative allogeneic stem cell transplantation provides effective therapy for patients with metastatic renal cell carcinoma. Based on the preliminary reports from other investigators treating patient with breast and ovarian cancer, the investigators of this study would propose treating an expanded cohort of patients with any metastatic solid tumor.

The principal endpoints of the trial will include incidence of durable engraftment, quality of hematopoietic and immune reconstitution, extent of donor chimerism, incidence and severity of acute and chronic graft versus host disease (GVHD), and incidence of long-term disease free survival (DFS). The investigators will evaluate the tumor response of patients with stable or progressive disease post-transplant to donor lymphocyte infusions (DLI). The investigators will also study the effects of DLI on T-cell immunity in the recipients.

DETAILED DESCRIPTION:
The trial is a pilot study in which patients with metastatic solid tumors will undergo non-myeloablative allogeneic hematopoietic stem cell transplantation. Patients whose immunosuppressive therapy has been tapered off, are without GVHD, and have evidence of residual or progressive disease will undergo DLI.

In recent years there have been attempts to harness the graft-versus-tumor effect of allogeneic bone marrow transplant to treat patients with metastatic solid tumors. Researchers at the NIH recently reported on 19 patients with refractory metastatic renal-cell carcinoma who had suitable donors and received a preparative regimen of cyclophosphamide and fludarabine followed by an infusion of a peripheral-blood stem-cell allograft from an HLA-identical sibling or a sibling with a mismatch of a single HLA antigen.49 They note that at the time of the last follow-up, 9 of the 19 patients were alive 287 to 831 days after transplantation (median follow-up: 402 days). Two had died of transplantation-related causes and 8 of progressive disease. In 10 patients (53%) metastatic disease regressed: 3 had a complete response, and 7 had a partial response. The patients who had a complete response remained in remission 27, 25, and 16 months after transplantation. Regression of metastases was delayed, occurring a median of 129 days after transplantation, and often followed the withdrawal of cyclosporine and the establishment of complete donor T-cell chimerism. They concluded that these results were consistent with a graft-versus-tumor effect and that non-myeloablative allogeneic stem cell transplantation can induce sustained regression of metastatic RCCA in patients who have had no response to conventional immunotherapy.

ELIGIBILITY:
Inclusion Criteria

Patients:

* Candidates for this trial will be patients with metastatic solid tumors for whom no standard therapy exists or who have evidence of measurable disease that is clearly progressing following standard biologic therapy or chemotherapy for metastatic disease.
* Patients must have a healthy family member who is HLA-identical to the recipient and who is willing and able to receive a course of G-CSF and undergo 2- 4 daily leukaphereses.
* Each patient must be willing to participate as a research subject and must sign an informed consent form.
* Patients must be ambulatory with good performance status (ECOG 0 or 1; Karnofsky PS 100-80%).
* Patients must have adequate organ function as defined by:

  1. WBC > 3000/mm3, plt > 100,000/mm3, and hemoglobin > 10gm/100ml
  2. Serum creatinine < 1.8mg/dl or Cr clearance > 60cc/min.
  3. Total bilirubin < 1.5mg/dl
  4. No evidence of congestive heart failure, symptoms of coronary artery disease, serious cardiac arrhythmias
  5. LVEF ≥40% by echocardiogram or MUGA scan (Patients whose LVEF is between 40% and 50% will have their cyclophosphamide dose reduced by 25% to 45 mg/kg/d for 2 days (total dose of 90 mg/kg).)
  6. FEV1 > 2.0 liters or > 75% of predicted for height and age.
* Patients must not be on systemic corticosteroids for intercurrent illness.
* Patients must be between 18 and 60 years of age. Patients over 60 will be accrued on an individual basis with approval of BMT service attendings.
* Women of childbearing potential must have a negative pregnancy test and not become pregnant while on treatment.

Donors:

* Absence of hematologic or marrow function-related diseases that interfere with the collection of sufficient numbers of normal progenitor cells.
* Absence of any medical condition that would pose a serious health risk to a patient undergoing peripheral blood stem cell harvest.
* Negative HIV, HTLV-1, and hepatitis C serologies.
* Negative for hepatitis B surface antigen (NOTE: Donors who are hepatitis B surface antibody and/or core antibody positive BUT hepatitis B surface antigen negative will be considered for transplant.)
* The donor must be a blood relation. Any healthy family member will be considered for marrow donation. Selection of a donor will be based on typing of HLA-A, B, DR loci to be carried out on the recipient, siblings, parents and possibly other family members such as aunts, uncles and cousins. A prospective related donor must be HLA identical to the patient.

Exclusion Criteria:

Patients:

* Patients with brain metastases, leptomeningeal disease or seizure. (NOTE: Patients with a history of brain metastases must be 6 months from definitive therapy (i.e. surgery or radiation) and have no evidence of disease or edema on brain CT scan or MRI.)
* Female patients who are pregnant or breast-feeding
* ECOG performance status >1. (Karnofsky PS <80%) (See Appendix 1.)
* Left ventricular ejection fraction of < 40%.
* Active viral (e.g. chronic active hepatitis), bacterial or fungal infection.
* Patients seropositive for HIV, HTLV -1,
* Patients not providing informed consent.
* Patients with known hypersensitivity to E. coli-derived products.

Donors:

* A positive HIV or HTLV-1 test or evidence of active/persistent viral hepatitis infection will exclude the donor from participation in this study. Donors who are HIV or HTLV-1 positive are ineligible because of the risk of transmission of virus during peripheral blood stem cell transplantation. Presence of any medical condition that would pose a serious health risk by undergoing peripheral blood stem cell harvest. Known hypersensitivity to E. coli-derived products.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2000-11; Primary Completion 2007-11 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine the percent 100-day survival of patients with metastatic solid tumors undergoing non-myeloablative allogeneic stem cell transplantation (SCT). | 100 days
To determine the incidence of treatment-related toxicity and acute and chronic graft versus host disease. | 100 days

SECONDARY OUTCOMES:
To determine the overall survival of patients with metastatic solid tumors undergoing non-myeloablative allogeneic SCT. | 2 years
To evaluate the tumor response in patients with metastatic solid tumors undergoing non-myeloablative allogeneic SCT. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David F McDermott, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States